CLINICAL TRIAL: NCT07377383
Title: Cardiometabolic Adaptations to Resistance and Endurance Exercise: Effects of Effort Configuration in Concurrent Training for Postmenopausal Women
Brief Title: Cardiometabolic Adaptations to Concurrent Training: Effect of Effort Configuration on Postmenopausal Women
Acronym: CARE+E
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade da Coruña (Other)
Collaborators: Ministerio de Ciencia, Innovación y Universidades, Spain (Unknown)
Responsible Party: Principal Investigator, Eliseo Iglesias Soler, Principal Investigator, Universidade da Coruña
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PID2024-156481OB-I00
Record Dates: First submitted 2025-12-24; First posted 2026-01-29 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Postmenopausal; Hypertension
Keywords: postmenopausal women; cardiovascular adaptations; concurrent training; resistance training; endurance training; interference phenomenon
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Short Set Configuration (4S) + Moderate-Intensity Continuous Training (MICT) (Experimental): Postmenopausal women perform a resistance training protocol with a Short Set Configuration (4 sets × 9 repetitions, 45 s inter-set rest, 4 min between exercises) and moderate-intensity continuous cycling (30 min at ~85% of anaerobic threshold).
  Interventions: Other: Concurrent Training Program
- Concurrent Training: Long Set Configuration (9S) + Moderate-Intensity Continuous Training (MICT) (Experimental): Postmenopausal women perform a resistance training protocol with a Long Set Configuration (9 sets × 4 repetitions, 120 s inter-set rest, 4 min between exercises) and moderate-intensity continuous cycling (30 min at ~85% of anaerobic threshold).
  Interventions: Other: Concurrent Training Program
- Concurrent Training: Short Set Configuration (4S) + Aerobic Interval Training, 30% TTE (AIT30) (Experimental): Postmenopausal women perform a resistance training protocol with a Short Set Configuration (4 sets × 9 repetitions, 45 s inter-set rest, 4 min between exercises) and aerobic interval training at low effort configuration (work intervals = 30% TTE, rest intervals adjusted to maintain work-to-rest ratio).
  Interventions: Other: Concurrent Training Program
- Concurrent Training: Long Set Configuration (9S) + Aerobic Interval Training, 30% TTE (AIT30) (Experimental): Postmenopausal women perform a resistance training protocol with a Long Set Configuration (9 sets × 4 repetitions, 120 s inter-set rest, 4 min between exercises) and aerobic interval training at low effort configuration (work intervals = 30% TTE, rest intervals adjusted to maintain work-to-rest ratio).
  Interventions: Other: Concurrent Training Program
- Concurrent Training: Short Set Configuration (4S) + Aerobic Interval Training, 75% TTE (AIT75) (Experimental): Postmenopausal women perform a resistance training protocol with a Short Set Configuration (4 sets × 9 repetitions, 45 s inter-set rest, 4 min between exercises) and aerobic interval training at high effort configuration (work intervals = 75% TTE, 1:1 work-to-rest ratio).
  Interventions: Other: Concurrent Training Program
- Concurrent Training: Long Set Configuration (9S) + Aerobic Interval Training, 75% TTE (AIT75) (Experimental): Postmenopausal women perform a resistance training protocol with a Long Set Configuration (9 sets × 4 repetitions, 120 s inter-set rest, 4 min between exercises) and aerobic interval training at high effort configuration (work intervals = 75% TTE, 1:1 work-to-rest ratio).
  Interventions: Other: Concurrent Training Program

INTERVENTIONS:
Other: Concurrent Training Program — All participants will follow a 20-week concurrent training program consisting of four supervised training sessions per week: two sessions of endurance training and two sessions of resistance training. Each resistance training session will include exercises targeting major muscle groups (leg press, bench press, prone leg curl, and lat pull-down). All exercises will be performed using the 12-repetition maximum load, completing a total of 36 repetitions per exercise. Inter-set rest periods will be arranged so that the total rest time per exercise is 6 minutes, maintaining a consistent work-to-rest ratio. Recovery between exercises will be 4 minutes. will consist of cycling exercises performed at prescribed intensities determined from incremental exercise testing. All sessions will have a total duration of thirty minutes. Work and recovery intervals will be arranged to maintain a consistent work-to-rest ratio across all participants.

SUMMARY:
The main objectives of this project are to assess the effects of a 20-week concurrent training program on neuromuscular adaptations, body composition, cardiometabolic health, quality of life, mood state, physical self-perception, and menopause-related symptoms in physically active postmenopausal women, and to compare the adaptations resulting from different combinations of endurance and resistance training programs with varying effort configurations.

Additionally, this project aims to examine the longitudinal interaction and potential interference effects between endurance and resistance training effort configurations throughout the training program and to determine the optimal combination of effort configurations that maximizes health benefits in concurrent training programs for physically active postmenopausal women.

DETAILED DESCRIPTION:
Menopause has a deleterious effect on women's health. The withdrawal of estrogens is associated with changes in body fat distribution, reduced glucose tolerance, abnormal lipid profiles, increased blood pressure, heightened sympathetic tone, endothelial dysfunction, and vascular inflammation. Training programs that combine endurance and resistance exercises-commonly referred to as concurrent training (CT) - at an optimal dose are recommended to counteract or even reverse some of the adverse effects of menopause.

This project builds upon a previous study conducted as part of a previous research project (PID2021-124277OB-I00), which examined the cardiovascular, metabolic, neuromuscular, and perceptual responses and adaptations of postmenopausal women to resistance training programs with different set configurations. The present proposal (CARE+E) extends this line of research by systematically incorporating the endurance component into CT programs and by manipulating effort configuration in both resistance and endurance exercises, thereby addressing a major limitation of the previous project, in which the cardiorespiratory training component was not experimentally controlled.

The inclusion of endurance training within a controlled CT framework enables the analysis of how resistance and endurance stimuli interact over time. In this context, the interference phenomenon, defined as the attenuation of adaptations induced by one exercise modality when it is combined with another within a concurrent training program, has been widely discussed but remains insufficiently understood, particularly with respect to the role of training load distribution. Effort configuration, defined as the duration of exercise sets relative to the maximal effort that can be sustained at a given intensity, may represent a key factor influencing this interaction. Nevertheless, the combined cardiometabolic and neuromuscular effects of different effort configurations in CT programs have not been systematically investigated, and evidence in physically active postmenopausal women is currently lacking.

By implementing a 20-week intervention, this project extends beyond the short- and medium-term durations typically used in postmenopausal populations, allowing for the evaluation of chronic adaptations to concurrent training. Periodic assessments throughout the program will provide insight into the longitudinal evolution of interactions between endurance and resistance training and will enable the identification of combinations of effort configurations that maximize health-related benefits. In this way, the project will generate novel evidence to inform the design of optimized concurrent training prescriptions tailored to the specific physiological characteristics of physically active postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* At least one year since the last menstrual period.
* Physically active, defined as engaging in 150-300 minutes of moderate physical activity per week or at least 75 minutes of vigorous activity per week.
* Three or fewer traditional cardiovascular risk factors.
* Asymptomatic and without cardiovascular (except controlled hypertension), metabolic, or renal diseases.
* In the case of hypertensive participants, well-controlled grade 1 hypertension managed with a single medication.

Exclusion Criteria:

* Diagnosis of grade 2 or grade 3 hypertension.
* Hypertension managed with more than one medication or with a drug that could interfere with cardiovascular responses to exercise (e.g., beta-blockers).
* Current or prior use of hormone replacement therapy.
* Hypertensive response to exercise.

Ages: 46 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Systolic, diastolic and mean blood pressure will be obtained by a photoplethysmography sensor. Units: mmHg
Baroreflex sensitivity | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Simultaneous electrocardiogram and beat-to-beat blood pressure recordings obtained by a photoplethysmography sensor will be used for calculating baroreflex sensitivity by sequential methods. Units: mmHg/ms
Heart rate variability in time domain | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Standard deviation of the normal-to-normal interval (SDNN) and root of the mean squared differences of successive NN intervals (RMSSD) will be obtained by analyzing inter-beat intervals from electrocardiogram recordings. Units: ms
Heart rate variability in frequency domain | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Obtained from spectral analysis of electrocardiogram recordings. High (HF) and Low (LF) frequency bands power will be determined by Fast Fourier Transformation method. Units: ms2/Hz
Blood pressure variability | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  It will be calculated by spectral analysis of beat-to-beat blood pressure recordings obtained by a photoplethysmography sensor. Units: mmHg2/Hz.
Arterial stiffness | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Pulse wave velocity will be measured at both the carotid-femoral and finger-toe segments. Units: m/s.
Resting metabolic rate | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  It will be obtained by measuring oxygen consumption at rest. Units: kcal/·day
Health-related quality of life (HRQoL) | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Health-Related Quality of Life assessed using the Cervantes Scale, which evaluates overall quality of life in postmenopausal women. The scale ranges from 0 to 100, with higher scores indicating better quality of life.
Menopause-Related Symptoms | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Menopause-Related Symptoms assessed using the Greene Climacteric Scale, which quantifies the severity and frequency of menopause symptoms. The scale ranges from 0 to 63, with higher scores indicating more severe menopause-related symptoms.
Mood State | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Mood State assessed using the Evaluation of Emotional States Mood Assessment Scale, which evaluates different dimensions of mood in participants. The scale ranges from 0 to 100, with higher scores indicating more positive mood.
Physical Self-Perception | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Physical Self-Perception assessed using the Physical Self-Perception Profile Scale, which evaluates body image and perceived physical competence. The scale ranges from 1 to 6, with higher scores indicating greater perceived physical competence and more positive body image.
Blood Lipid Profile | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Biochemical variables related to dyslipidemia, including total cholesterol, LDL, HDL, and triglycerides, measured using a portable cholesterol analyzer (ACON Laboratories, USA).
Blood Glucose | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Fasting Blood Glucose measured in milligrams per deciliter using a multiparameter monitor (Gimacare, Gima S.P.A., Italy).
Oxidative Stress Markers (Total Antioxidant Capacity) | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Total Antioxidant Capacity measured in millimoles of Trolox equivalents per liter using the BRS-BQC Redox System (BQC Redox Technologies, Spain).
Power-velocity relationship | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Relationship betweenPower (W) and angular velocity (°/s). Obtained by performing maximum torque at specific velocities in an isokinetic dynamometer
Maximum isometric torque | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Maximum torque recorded at fixed angular position. It will be measured with an isokinetic dynamometer. Units: N/m
Hemoglobin | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Hemoglobin concentration measured in grams per deciliter using a multiparameter monitor (Gimacare, Gima S.P.A., Italy).
Oxidative Stress Markers (Hydrogen Peroxide Scavenging Capacit) | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Hydrogen Peroxide Scavenging Capacity measured in micromoles per liter using the BRS-BQC Redox System (BQC Redox Technologies, Spain).

SECONDARY OUTCOMES:
Physical Activity Level | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Physical Activity Level assessed using the International Physical Activity Questionnaire, which evaluates walking, moderate-intensity, and vigorous-intensity activities performed in a typical week across all domains of daily life, including leisure time activities, domestic and gardening activities, work-related activities, and transport activities.
  Participants are classified into three categories: Inactive (not meeting the criteria for minimally active or health-enhancing physical activity active), Minimally Active (achieving at least six hundred metabolic equivalent minutes per week through a combination of activity types), and Health-Enhancing Physical Activity Active (exceeding the minimum recommended levels of physical activity for health). Higher categories indicate greater habitual physical activity and better adherence to public health recommendations.
Dietary Habits | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Assessed using the Short Diet Quality Screener (SDQS) questionnaire to evaluate dietary patterns and quality.
Body Composition: Body Fat Percentage | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Body Fat Percentage measured in percent using multifrequency bioimpedance (Bodystat Quadscan 4000, Quadscan, United Kingdom).
Bone Mineral Density | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Estimated bone mineral density assessed using ultrasound densitometry (Sonost 3000, Osteosys Corp., Korea).
Muscle Morphology | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Muscle thickness and cross-sectional area of biceps brachii and vastus lateralis measured by ultrasound (Versana Active device with 12L-RS linear probe, GE HealthCare, USA).
Cardiorespiratory Fitness (Peak oxygen uptake) | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Peak Oxygen Uptake, in order to asses the cardiorespirtoty fitness, measured in milliliters per kilogram per minute during an incremental cycle ergometer test.
Time to Exhaustion (TTE) | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Duration (in seconds or minutes) that participants maintain a power output corresponding to 90% of VO₂max at a cadence of 75-85 rpm during a constant-load cycling test.
Balance | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Postural stability measured by center of pressure displacement during the Romberg test using a force platform (Kistler Instrumente AG, Switzerland).
Muscular Strength | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Assessed using the 12RM load for each resistance exercise, with execution velocity recorded to evaluate the loss of propulsive velocity during repetitions.
Body Composition: Lean Mass | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Lean Mass measured in kilograms using multifrequency bioimpedance (Bodystat Quadscan 4000, Quadscan, United Kingdom).
Body Composition: Total Body Water | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Total Body Water measured in liters using multifrequency bioimpedance (Bodystat Quadscan 4000, Quadscan, United Kingdom).
Exercise Heart Rate | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Heart Rate measured in beats per minute during an incremental cycle ergometer test.
Exercise Blood Pressure | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Systolic nad Diastolic Blood Pressure measured in millimeters of mercury during an incremental cycle ergometer test.
Individualized Power Output | Baseline (week 0), partial evaluation 1 (week 6), partial evaluation 2 (week 12), partial evaluation 3 (week 18), and post-intervention evaluation (week 24)
  Individualized Power Output measured in watts, determined from the regression between external load and percentage of maximal oxygen uptake during an incremental cycle ergometer test.

OTHER OUTCOMES:
Health Status | Baseline (week 0)
  Assessed by a medical professional during the preliminary consultation using standard clinical evaluation procedures.
Cardiovascular Risk Factors | Baseline (week 0)
  Stratified during the preliminary medical consultation. Participants will be categorized into standardized cardiovascular risk levels (for example, low risk, moderate risk, or high risk) according to established clinical criteria that combine blood pressure category (e.g., high-normal, Grade 1 hypertension, Grade 2 hypertension) with the number of additional risk factors and presence of organ damage or prior cardiovascular disease; higher categories indicate greater cardiovascular risk.
Absolute and Relative Contraindications for Exercise | Baseline (week 0)
  Assessed by a medical professional during the preliminary consultation using established clinical guidelines.
Resting Electrocardiogram Parameters | Baseline (week 0)
  Measured in standard clinical units during a resting electrocardiogram.
Resting Spirometry Measurements | Baseline (week 0)
  Measured in liters during a resting spirometry test, including forced vital capacity and forced expiratory volume in one second.

CONTACTS AND LOCATIONS:
Overall Officials: Eliseo Iglesias-Soler, PhD, Principal Investigator — Universidade da Coruña; María Rúa-Alonso, PhD, Principal Investigator — Universidade da Coruña

IPD SHARING:
Plan to Share IPD: Yes
After finishing the protocols (six months approximately) main data will be shared through European data repository Zenodo, in which University of A Coruna has created a community
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after finishing the whole project